CLINICAL TRIAL: NCT01801969
Title: Return to Work and QOL Following TBI. Impact of Rehabilitation Service.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: hovedtraume
Record Dates: First submitted 2013-02-06; First posted 2013-03-01 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Brain Injuries; Return to Work; Quality of Life
Keywords: Brain injuries; Rehabilitation services; Return to Work; Quality of life
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rehabilitation service: * Centralized or Decentralized rehabilitation
  * Size of municipality
  Interventions: Other: Rehabilitation service

INTERVENTIONS:
Other: Rehabilitation service — * Centralized/ decentralized hospital based rehabilitation defined as hospital based rehabilitation in a single or in multiple locations, respectively.
  * Size of the municipality responsible for providing rehabilitation services after discharge from hospital

SUMMARY:
The proportion of patients who return to work after surviving severe traumatic brain injury (TBI) has been estimated in number of studies but results do not agree.This may be due to complex interaction between many factors, including available rehabilitation services.

In Denmark rehabilitation services vary been regions and municipalities. Hospital based rehabilitation is organized by the regions. Rehabilitation outside the hospitals is organized by the municipalities

The first purpose of this study is to investigate a possible link between centralized hospital based rehabilitation and better return to work / quality of life.

The second purpose is to investigate whether municipality size affects quality of life and return to work after severe TBI.

Data on return to work are derived from a national register on labor market attachment. Data on quality of life are derived from a questionnaire.

The study population is identified from the Danish Head Trauma Database. The completeness and accuracy of the database will be investigated as the first part of the project.

ELIGIBILITY:
Inclusion Criteria:

* age 18-64

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals suffering from severe TBI (GCS<9) from the Danish Head Trauma Database
Sampling Method: Non-Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
time to return to work | up to 11 years post-injury
  Data Source: Register (DREAM)

SECONDARY OUTCOMES:
Quality of life | 1-10 years post-injury
  Data Source: Questionnaire (QUOLIBRI)

CONTACTS AND LOCATIONS:
Overall Officials: Lene Odgaard, Principal Investigator — Research Unit (Forskningsenheden), Hammel Neurorehabilitation and Research Centre
Locations (1):
- Hammel Neurorehabilitation and Research Centre, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No